CLINICAL TRIAL: NCT03510247
Title: What Physiological Changes Occur During the Competitive Rugby Union Season?
Brief Title: Physiological Changes Throughout the Competitive Rugby Season.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Surrey (Other)
Responsible Party: Principal Investigator, Victoria Benford, Principal Investigator, University of Surrey
Other Study IDs: UoS-Quins1
Record Dates: First submitted 2018-04-17; First posted 2018-04-27 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Body Composition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rugby union is a high intensity, intermittent team sport which is played over 80 minutes. Players are divided into two main positional groups, forwards and backs, with backs covering a larger distance and completing more sprints and forwards partaking in more static exertions. With the game of rugby union getting progressively faster, body composition and power to weight ratio are key determinants. Due to the demands placed on these players it is essential that they are in optimal health continually, however, whilst the required physical attributes are well documented, this research will provide an insight into physiological and anthropometric changes that occur across two seasons.

During this study subjects will be asked to attend the lab on 8 occasions over the course of two seasons (June 2018, September 2018, January 2019, April 2019, June 2019, September 2019, January 2020 and April 2020). During these visits the following tests will be completed; a peripheral Quantitative Computed Tomography (pQCT) scan of the bone mineral composition of the tibia and radius, total body composition via Dual Energy X-ray Absorptiometry (DXA), anterior-posterior spine bone mineral density to assess fracture risk via DXA, vertebral fracture risk via DXA. ~24ml of whole blood will be taken to determine serum 25(OH)D, albumin, calcium, zinc, total red blood cell count, lymphocytes, monocytes, carboxy-terminal collagen crosslinks (CTX) and amino-terminal propeptide (P1NP) concentrations. In June all players will complete a 6 minute run to determine fitness. Players will be expected to measure body weight and complete wellness questionnaires daily at the club and have skinfold measurements taken monthly. global positioning system (GPS) data will be collected during each training session and performance analysis will be utilised to determine the amount of contacts completed. Illness and injury occurrences will be recorded throughout the season.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18-35 years old
* Contracted player of Harlequins Rugby Club

Exclusion Criteria:

* Any participant who has been exposed to radiation exceeding 5millisieverts within the past 12 months will be excluded from dual-energy X-ray absorptiometry (DXA) and peripheral quantitative computed tomography (pQCT) scans for the relevant time points, however all other (non-ionizing) measures will be collected.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Male elite rugby union players.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2018-05 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Fat percentage | Two years
  Body fat percentage (%) change over the course of two seasons.
Muscle Mass | Two years.
  Total muscle mass (kg) change over the course of two seasons

SECONDARY OUTCOMES:
Fracture Risk | Two Years
  Bone mineral density, vertebral fracture assessment and bone structure will be combined to determine fracture risk over the course of two seasons.
Vitamin D Status | Two years
  Vitamin D status (25(OH)D) will be measured over two seasons to determine seasonal changes.